CLINICAL TRIAL: NCT06201858
Title: Examining Engagement Trends Among Participants in Hidradenitis Suppurativa Clinical Trials
Brief Title: A Journey Into Participation Patterns Among Patients With Hidradenitis Suppurativa
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 67172350
Record Dates: First submitted 2023-12-29; First posted 2024-01-11 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to uncover the factors driving patient decisions regarding enrollment, withdrawal, or re-engagement in hidradenitis suppurativa clinical trials. Understanding these factors will significantly improve the relevance and effectiveness of future research endeavors.

Ultimately, this trial endeavors to deepen our understanding of the factors impacting hidradenitis suppurativa clinical trial participation. Enhancing participation rates could accelerate the development of innovative treatments for this debilitating condition.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old
* Diagnosis of hidradenitis suppurativa
* Able to comprehend the investigational nature of the protocol and provide informed consent

Exclusion Criteria:

* Female patients who are currently pregnant or nursing
* Inability to perform regular electronic reporting
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hidradenitis suppurativa who are actively considering enrolling in a clinical study for said condition, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Number of hidradenitis suppurativa patients who decide to enroll in a clinical research | 3 months
Rate of hidradenitis suppurativa patients who remain in clinical trial to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Saunte DML, Jemec GBE. Hidradenitis Suppurativa: Advances in Diagnosis and Treatment. JAMA. 2017 Nov 28;318(20):2019-2032. doi: 10.1001/jama.2017.16691. PMID 29183082
- [Background] Garcovich S, Fania L, Caposiena D, Giovanardi G, Chiricozzi A, De Simone C, Tartaglia C, Ciccone D, Bianchi L, Abeni D, Peris K. Pediatric Hidradenitis Suppurativa: A Cross-Sectional Study on Clinical Features and Treatment Approaches. J Cutan Med Surg. 2022 Mar-Apr;26(2):127-134. doi: 10.1177/12034754211039993. Epub 2021 Oct 6. PMID 34615396
- [Background] Jfri A, Nassim D, O'Brien E, Gulliver W, Nikolakis G, Zouboulis CC. Prevalence of Hidradenitis Suppurativa: A Systematic Review and Meta-regression Analysis. JAMA Dermatol. 2021 Aug 1;157(8):924-931. doi: 10.1001/jamadermatol.2021.1677. PMID 34037678

DOCUMENTS (1):
  • Informed Consent Form (2023-12-29): https://cdn.clinicaltrials.gov/large-docs/58/NCT06201858/ICF_000.pdf